CLINICAL TRIAL: NCT04649944
Title: Assessment of the Serological Profile of Children and Adolescents Between 4 and 16 Years of Age Cohabiting With at Least One Family Member Who Tested Positive to COVID-19: an Observational Study
Brief Title: Serological Profile of Children and Young Adolescents With at Least One COVID-19 Diagnosed Family Member
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Marco Farronato, Principal Investigator, University of Milan
Other Study IDs: GMT_CD_CT_LG_EB_10_2020
Record Dates: First submitted 2020-11-26; First posted 2020-12-02 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: Sars-Cov-2; serological test; children; young adults; positive naso-pharyngeal swab; family cluster
MeSH Terms: conditions — COVID-19 | interventions — Serologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will collect blood samples from subjects' finger
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serological test and phone interview — Families are interviewed by telephone to gather information about the family cluster (i.e. age and number of cohabitants, their symptoms and swab results, if performed), the subject who tested positive (i.e.sex, age, course of the disease, symptoms suggestive of COVID-19) and children aged between 4 and 16 y.o. (i.e. sex, age, drug therapy and/or chronic diseases, symptoms suggestive of COVID-19).
  Children, young adults and the cohabitant who previously tested positive to the swab undergo a serological test for the detection of IgG and IgM antibodies for Sars-Cov-2.

SUMMARY:
Use of rapid serological tests to assess the vulnerability to SARS-CoV-2 infection of subjects aged 4-16 years old and cohabiting with at least one family member who tested positive to SARS-CoV-2

DETAILED DESCRIPTION:
Families with at least one child or young adult aged between 4 and 16 years old and with at least one cohabitant who tested positive to nasopharyngeal swab are contacted by phone. Those who decide to sign an informed consent after reading the study information will be included in the study. It consists of a preliminary telephone interview and a following rapid serological test for all children and young adults with the age included in the range of interest and the cohabitant who tested positive to nasopharingeal swab.

The obtained results will be collected and analysed, and the outcomes of the study will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Children and young adults aged between 4 and 16 years old with at least a Sars-Cov-2 positive cohabitant
2. Adults who previously tested positive to SARS-CoV-2 with at least a cohabitant aged between 4 and 16 y.o.
3. Subjects from the district of Sesto San Giovanni, Lombardy, Italy

Exclusion Criteria:

1. Children and young adults aged between 4 and 16 years old without at least a cohabitant who previously tested positive to SARS-CoV-2
2. Adults who previously tested positive to SARS-CoV-2 without at least a cohabitant aged between 4 and 16 y.o.
3. Absence of a signed informed consent
4. Subject with symptoms suggestive of COVID-19 in the last 14 days or disease in progress

Ages: 4 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and young adults aged between 4 and 16 years old, both males and females, with at least a cohabitant who previously tested positive to SARS-CoV-2 Adults who previously tested positive to SARS-CoV-2, both males and females, with at least a cohabitant aged between 4 and 16 y.o.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-02-05 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of IgG and IgM antibodies for Sars-Cov-2 in children aged between 4 and 16 y.o. cohabiting with at least a subject with a previous diagnosis of COVID-19. | 1-30 days
  Assessment of IgG and IgM using serological tests at a single time point.

SECONDARY OUTCOMES:
Detection of IgG and IgM antibodies for Sars-Cov-2 in adults with a previous diagnosis of COVID-19 cohabiting with at least a child aged between 4 and 16 y.o. | 1-30 days
  Assessment of IgG and IgM using serological tests at a single time point.

CONTACTS AND LOCATIONS:
Overall Officials: Giampietro Farronato, DDS, Study Director — University of Milan
Locations (1):
- UOC Maxillofacial Surgery and Odontology, University of Milan, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
IPD are not planned to be available

REFERENCES:
- [Background] Ludvigsson JF. Systematic review of COVID-19 in children shows milder cases and a better prognosis than adults. Acta Paediatr. 2020 Jun;109(6):1088-1095. doi: 10.1111/apa.15270. Epub 2020 Apr 14. PMID 32202343
- [Background] Saleem H, Rahman J, Aslam N, Murtazaliev S, Khan S. Coronavirus Disease 2019 (COVID-19) in Children: Vulnerable or Spared? A Systematic Review. Cureus. 2020 May 20;12(5):e8207. doi: 10.7759/cureus.8207. PMID 32577325
- [Background] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261
- [Background] Sun D, Zhu F, Wang C, Wu J, Liu J, Chen X, Liu Z, Wu Z, Lu X, Ma J, Peng H, Xiao H. Children Infected With SARS-CoV-2 From Family Clusters. Front Pediatr. 2020 Jun 23;8:386. doi: 10.3389/fped.2020.00386. eCollection 2020. PMID 32656172